CLINICAL TRIAL: NCT05514834
Title: Feasibility Study to Evaluate the Safety and Efficacy of Cellular MAtrix™ BCT-HA Kit as a New Treatment Option for Dehydrated and Wrinkled Skin (A Clinical and Histological Evaluation)
Brief Title: BCT-HA Kit for Dehydrated and Wrinkled Skin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DERM-2021-30292
Record Dates: First submitted 2022-07-25; First posted 2022-08-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Rhytides; Wrinkle
Keywords: rhytides; wrinkles; facial aging; PRP; hyaluronic acid

STUDY DESIGN:
Intervention Model Description: Blinded, randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, and dermatopathologist (outcomes assessor) will all be blinded to which group the participant belongs too. Given the color difference of the injected solutions, the syringes with the injection material (HA with PRP or saline) will be masked to prevent the patient or investigator from knowing which material they are injecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- combined HA with PRP (Experimental): Hyaluronic acid and PRP combination treatment
  Interventions: Device: Cellular Matrix TM BCT-HA Kit (ref. BCT-HA-3)
- Placebo (Placebo Comparator): saline solution
  Interventions: Other: Placebo
- PRP (Active Comparator): Platelet rich plasma without hyaluronic acid
  Interventions: Other: PRP Only

INTERVENTIONS:
Device: Cellular Matrix TM BCT-HA Kit (ref. BCT-HA-3) — Injections with platelet-rich plasma and hyaluronic acid
  Arms: combined HA with PRP
Other: PRP Only — platelet rich plasma without hyaluronic acid
  Arms: PRP
Other: Placebo — Neither PRP nor hyaluronic acid
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of Cellular MatrixTM BCT-HA Kit treatment compared to placebo condition on revitalization and skin rejuvenation on the midface. Particular attention will be made to the safety aspects, as well as the histological consequences of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPPA Authorization
* Healthy men and women, ages 30 - 65 years of age
* Subjects with Fitzpatrick photo skin type I-VI
* Subjects with moderate to severe nasolabial folds contour deficiencies or other facial wrinkles. Degree of nasolabial folds or other facial wrinkles will be determined on the basis of the Wrinkles Severity Rating Scale
* Subjects who agree not to have any other procedures of affecting skin quality (microdermabrasion, peels, acne treatments, toxin, fillers etc.) for the duration of the study
* Subjects who understand the study and are able to follow study instructions and are willing to attend the required study visits.
* Subjects who agree to be photographed for research purposes and their identity may not be concealed in these photographs.

Exclusion Criteria:

* Subjects who have had any kind of aesthetic therapy (peeling, laser, ultrasound, toxins, fillers) in the facial area during the last 6 months
* Presence of implant in the facial area to treat
* Contraindications to the use of antiseptics (Biseptine, Amukine)
* Subjects who have an active or known skin inflammation or infection within the treatment area.
* Subjects who have an active or known acute skin allergies
* Subjects who have a known allergy to hyaluronic acid
* Subjects who have any other dermatologic conditions including acne, rosacea, eczema, psoriasis, actinic keratosis, severe sun damage, infection, or scars within the treatment area.
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy, or bilateral oophorectomy.
* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy.
* Subjects who have been diagnosed with diabetes
* Subjects who are Immunosuppressed
* Subjects who are HIV+ / VHB+ / VHC+
* Subjects who have had/will have a COVID vaccine within 2 weeks of study participation
* Subjects who have had/will have a dental procedure within 4 weeks of study participation
* Subjects with a history of severe bee allergy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Skin Quality Rating Scale | Week 32
  Skin Quality Rating Scale is a 10 point scales used to assess skin quality, including radiance, smoothness, pigmentation, erythema, and pore size.
Change in Global Aesthetic Improvement Scale | Week 32
  This is a 7 point scale to assess degree of improvement of facial skin after treatment.
Change in FACE-Q Score | Week 32
  The following eight FACE-Q scales: (1) satisfaction with overall facial appearance (measures patient satisfaction with the overall appearance of their face); (2) satisfaction with decision (measures patient satisfaction with their decision to undergo the procedure;(3) cheekbones; (4) chin; (5) cheeks; (6) lower face; (7) jawline; and (8) nasolabial folds (items 3 through 8 measure overall and area-specific appearance appraisal to evaluate satisfaction with specific facial areas). Higher FACE-Q scores indicate superior satisfaction
Physician's Global assessment to measure quality of life | 4 weeks after treatment 1st, 2nd and 3rd treatments and 32 weeks after enrollment
  Patient rating of improvement in treated area ranging from 1 to 5, with 5 being worse.
Visual Analog Score for patients | Immediately after 1st, 2nd and 3rd treatments
  Visual analog rating of pain associated with treatment administration ranging between 0 and 10, pain scale.
Wrinkle assessment | Week 32
  Wrinkle Assessment Score is a 9 point scale to asses severity of wrinkles.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States